CLINICAL TRIAL: NCT06554366
Title: Bacterial Load Reduction by GentleWave and EdgePro Irrigation Systems in Mandibular Necrotic Molars: An In-vivo Study
Brief Title: Bacterial Load Reduction by GentleWave and EdgePro Irrigation Systems in Mandibular Necrotic Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, David E Jaramillo, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-24-0062
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pulp Necroses
Keywords: Root canal
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- GentleWave (Experimental)
  Interventions: Device: GentleWave
- EdgePro (Experimental)
  Interventions: Device: EdgePro laser irrigation
- Irrisafe passive ultrasonic irrigation (Active Comparator)
  Interventions: Device: Irrisafe passive ultrasonic irrigation

INTERVENTIONS:
Device: GentleWave — Root canals will be shaped using a Vortex Blue and ProTaper gold rotary system. Once the root canals have been shaped, the GentleWave procedure will be performed
  Arms: GentleWave
Device: EdgePro laser irrigation — Root canals will be shaped using a Vortex Blue and ProTaper gold rotary system. Once the root canals have been shaped, the EdgePro procedure will be performed
  Arms: EdgePro
Device: Irrisafe passive ultrasonic irrigation — Root canals will be shaped using a Vortex Blue and ProTaper gold rotary system. Once the root canals have been shaped, the passive ultrasonic irrigation procedure will be performed
  Arms: Irrisafe passive ultrasonic irrigation

SUMMARY:
The purpose of this study is to compare the efficacy of GentleWave versus EdgePro irrigation in the disinfection of infected root canals of human permanent teeth with necrotic pulp.

ELIGIBILITY:
Inclusion Criteria:

* Permanent teeth that are diagnosed with pulp necrosis.
* elected to have a permanent tooth nonsurgical root canal treatment
* Signed informed consent.

Exclusion Criteria:

* Teeth with root fractures or previously root canal treated teeth.
* Teeth with severe loss of structure
* Teeth with vital pulps.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Bacterial count reduction checked by 16 S rDNA next-generation sequencing analysis (NGS) | Baseline, after cleaning and shaping of the root canal (about 30 minutes after baseline)

SECONDARY OUTCOMES:
Presence of proteolytic versus non-proteolytic bacteria in the root canals | Baseline, after cleaning and shaping of the root canal (about 30 minutes after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: David Jaramillo, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No